CLINICAL TRIAL: NCT04228744
Title: Deep Brain Stimulation for Refractory Obsessive-Compulsive Disorder: Efficacy and Mechanism of Ventral Internal Capsue and Nucleus Accumbens
Brief Title: The Efficacy and Mechanism of DBS in VIC and NAcc for Refractory OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of Functional Neurosurgery Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019 NAc VIC DBS OCD
Record Dates: First submitted 2020-01-05; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Obsessive-Compulsive Disorder; Deep Brain Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral surgical implantation of DBS system (Experimental): All the participants will receive bilateral surgical implantation of DBS system to VIC and NAc. The experimenter will active the DBS system and adjust the parameters for all the participants after surgery.
  Interventions: Device: DBS system

INTERVENTIONS:
Device: DBS system — The DBS device utilized in the present study includes a dual-channel neurostimulator kit, lead kit, extension kit, clinician-operated wireless programmer, test stimulator, and patient controller. The lead contains four stimulating contacts. The length of each contact is 1.5 mm, and the spacing between contacts is 1.5 mm.
  The participants will receive stepwise surgery. The electrodes will be implanted firstly which will be externalized for several days and then the IPG will be implanted. During externalization, the experimenters will record the local field potential and electroencephalography in resting or task-based state with conditions of sham-stimulation or active-stimulation.

SUMMARY:
This study will evaluate the efficacy and explore the mechanism of deep brain stimulation (DBS) in the ventral internal capsule (VIC) and nucleus accumbens (NAc) for refractory obsessive-compulsive disorder (OCD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OCD with duration of at least 5 years;
2. Severity rated as severe to extreme illness;
3. Failed adequate trial of at least three specific serotonin reuptake inhibitor (SSRI) antidepressants;
4. Failed augmentation with antipsychotic;
5. Completed or failed to complete adequate trial of cognitive behavioural therapy for OCD;
6. Stable medication regimen for one month before surgery;
7. Signed informed consent;

Exclusion Criteria:

1. Hoarding as a primary symptom;
2. No other serious psychiatric disorder such as psychotic disorder;
3. Drug or substance use disorder within 6 months except nicotine;
4. Major Neurological/Medical condition;
5. High suicide risk;
6. Pregnancy or lactation;
7. Contraindications to stereotactic surgery;
8. Contraindications to MRI;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  Y-BOCS is used to rate the severity of OCD symptoms by clinicians. Higher score means more severe OCD symptoms.

SECONDARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale-Self Report (Y-BOCS-SR) Score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The Y-BOCS-SR is a self-report version of the clinician-rated Y-BOCS. It consists of 10 items rated on a 5-point Likert scale (0 to 4) with higher scores denoting greater symptom severity.
Change in Yale-Brown Obsessive-Compulsive Scale-Second Edition (Y-BOCS-II) Score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The Y-BOCS-II was created given several overarching concerns about the original Y-BOCS. Each item is rated from 0 to 5, and higher score means more severe OCD symptoms.
Change in Obsessive-Compulsive Inventory - Revised (OCI-R) Score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The OCI-R is an 18-item self-reported scale that assesses the degree of distress caused by OCD symptoms. Each item is rated from "not at all" (codes as 0) to "extremely" (codes as 4), and three items constitute a subtype of OCD symptoms.
Adverse Events | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
Changes in Hamilton Anxiety Scale Score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The Hamilton Anxiety Scale is a clinician-rated scale. Higher scores indicate more severe anxiety.
Changes in Hamilton Depression Scale-17 Score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The Hamilton Depression Scale-17 is a clinician-rated scale. Higher scores indicate more severe depression.
Magnetic resonance imaging (MRI) images | Baseline (preoperative)
  The MRI images contains resting, multi-tasks related, and structural states.
Change in memory | Baseline (preoperative),6 months or 12 months
  The CANTAB software research is used to assess memory and learning. The tasks incude spatial working memory task, paired associated learning task, pattern recognition memory task.
Change in impulsivity and compulsivity | Baseline (preoperative),6 months or 12 months
  The computerized tasks are used to measure impulsivity and compulsivity. The tasks include stop single task, beads task, model-based modle-free task and habit task.
Change in Young Manic Rating Scale(YMRS) | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The YMRS is a 11-item rating scale used to evaluate manic symptoms. Higher score indicates more severe mania.
Changes in SF-36 score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The 36-Item Short Form Survey (SF-36) is used to measure the quality of life. The higher score means higher quality of life.
Changes in WHOQOL-BREF score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The WHOQOL-BREF is used to measure the quality of life. The higher score means higher quality of life.
Changes in Q-LES-Q-SF score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The quality of life enjoyment and satisfaction questionnaire - short form (Q-LES-Q-SF) is used to measure the quality of life. The higher score means higher quality of life.
Changes in PSQI score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The pittsburgh sleep quality index (PSQI) is used to measure the quality and patterns of sleep. Higher score means poorer quality of sleep.
Changes in PSS-10 score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The perceived stress scale (PSS-10) is used to measure stress levels and contains 10 items rated from "never" (coded as 0) to "very often" (coded as 4). Higher score means higher level of stress.
Changes in PANAS score | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The positive and negative affective schedule (PANAS) consists of 20 words that describe different feeling and emotions. 10 words constitute negative affect and positive affect subscales. Each word was rated from "very slightly or not at all" (coded as 1) to "extremely" (coded as 5). Higher score means higher level of positive or negative affect.
Change in Sheehan Disability Scale | Baseline (preoperative), 1 month, 3 months, 6 months, 12 months, 18 months
  The Sheehan Disability Scale is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired. The patient rates the extent to which his or her 1) work, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine; Valerie Voon, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Ruijin Hospital, Shanghai, China